CLINICAL TRIAL: NCT05088811
Title: The Role of Long Non-coding RNAs WRAP53 and UCA-1 as Potential Biomarkers in Diagnosis of Hepatocellular Carcinoma
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Alexandria University (Other)
Responsible Party: Principal Investigator, Elsheaita, Ahmed Mohamed Elmoughazy Abdelfatah Aly, Assistant lecturer, experimental and clinical internal medicine, medical research institute, Alexandria University
Other Study IDs: HCC medical research institute
Record Dates: First submitted 2021-08-21; First posted 2021-10-22 (Actual); Last update posted 2021-10-22 (Actual); Status verified 2021-10

CONDITIONS: Hepatocellular Carcinoma; Liver Cirrhosis; Diagnoses Disease
Keywords: Hcc, liver cirrhosis, UCA-1, WRAP53
MeSH Terms: conditions — Carcinoma, Hepatocellular; Liver Cirrhosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Serum specimen
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Liver cirrhosis: Group (1): Thirty patients having liver cirrhosis and hepatocellular carcinoma diagnosed by tripahsic CT.
  Interventions: Diagnostic Test: WRAP53, UCA-1
- Hepatocellular Carcinoma: Group (2): Thirty liver cirrhosis patients without hepatocellular carcinoma diagnosed by abdominal ultrasound examination
  Interventions: Diagnostic Test: WRAP53, UCA-1
- Control: Group (3): Twenty normal subjects (control group) matching in age and sex with patients in groups 1 and 2.
  Interventions: Diagnostic Test: WRAP53, UCA-1

INTERVENTIONS:
Diagnostic Test: WRAP53, UCA-1 — Diagnostic value of UCA-1 and WRAP53 in HCC

SUMMARY:
The aim of this work is to study the role of long non-coding RNAs WRAP53 and urothelial carcinoma-associated 1 (UCA1) as potential biomarkers in diagnosis of hepatocellular carcinoma.

DETAILED DESCRIPTION:
Sample size calculation was done in department of medical statistics, Medical Research Institute, Alexandria University and the total minimal sample size was calculated.

A prospective case control study will be conducted on 80 subjects divided into three groups:

Group (1): Thirty patients having liver cirrhosis and hepatocellular carcinoma diagnosed by tripahsic CT.

Group (2): Thirty liver cirrhosis patients without hepatocellular carcinoma diagnosed by abdominal ultrasound examination.

Group (3): Twenty normal subjects (control group) matching in age and sex with patients in groups 1 and 2.

Patients will be recruited from the outpatient clinics and inpatient wards of Alexandria Main University Hospital and Medical Research Institute Hospital. Full informed consent will be taken from the patients and approval of the ethical committee of the Faculty of Medicine will be fulfilled. Exclusion criteria: Patients with any inflammatory diseases or other malignancies.

ELIGIBILITY:
Inclusion Criteria:

* Any subject without any of the exclusion criteria

Exclusion Criteria:

* Patients with any inflammatory diseases or other malignancies.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Group (1): Thirty patients having liver cirrhosis and hepatocellular carcinoma diagnosed by tripahsic CT.
  Group (2): Thirty liver cirrhosis patients without hepatocellular carcinoma diagnosed by abdominal ultrasound examination.
  Group (3): Twenty normal subjects (control group) matching in age and sex with patients in groups 1 and 2.
Sampling Method: Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2021-08-21 (Actual); Primary Completion 2022-08 (Estimated); Study Completion 2022-09 (Estimated)

PRIMARY OUTCOMES:
Diagnostic value of long non coding RNA UCA-1 and WRAP53 in Hepatolcellular carcinoma | One year
  Calculating sensitivity and specifity of UCA-1 and WRAP53 to assess their diagnostic value in diagnosis of hepatocellular carcinoma

CONTACTS AND LOCATIONS:
Locations (2):
- Egypt (2):
  - Alexandria University, faculty of medicine, Alexandria
  - Alexandria University, medical research institute, Alexandria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Kamel MM, Matboli M, Sallam M, Montasser IF, Saad AS, El-Tawdi AHF. Investigation of long noncoding RNAs expression profile as potential serum biomarkers in patients with hepatocellular carcinoma. Transl Res. 2016 Feb;168:134-145. doi: 10.1016/j.trsl.2015.10.002. Epub 2015 Oct 24. PMID 26551349
- [Result] Pouladi N, Abdolahi S, Farajzadeh D, Hosseinpour Feizi MA. Haplotype and linkage disequilibrium of TP53-WRAP53 locus in Iranian-Azeri women with breast cancer. PLoS One. 2019 Aug 6;14(8):e0220727. doi: 10.1371/journal.pone.0220727. eCollection 2019. PMID 31387111
- [Result] Wang F, Ying HQ, He BS, Pan YQ, Deng QW, Sun HL, Chen J, Liu X, Wang SK. Upregulated lncRNA-UCA1 contributes to progression of hepatocellular carcinoma through inhibition of miR-216b and activation of FGFR1/ERK signaling pathway. Oncotarget. 2015 Apr 10;6(10):7899-917. doi: 10.18632/oncotarget.3219. PMID 25760077
- [Derived] Abdelmoety AA, Elhassafy MY, Said RSO, Elsheaita A, Mahmoud MM. The role of UCA1 and WRAP53 in diagnosis of hepatocellular carcinoma: A single-center case-control study. Clin Exp Hepatol. 2023 Jun;9(2):129-137. doi: 10.5114/ceh.2023.127569. Epub 2023 Jun 18. PMID 37502440